CLINICAL TRIAL: NCT01840605
Title: A Confirmatory Study of TAU-284 in Pediatric Patients With Atopic Dermatitis (Ketotifen Fumarate-controlled, Double-blind, Comparative Study)
Brief Title: A Confirmatory Study of TAU-284 in Pediatric Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAU-284-19
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Dermatitis; Atopic
MeSH Terms: conditions — Dermatitis | interventions — bepotastine besilate; Ketotifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAU-284 (Experimental): Two TAU-284 5mg tablets and one ketotifen fumarate dry syrup 1g placebo will be taken orally twice a day, once after breakfast and once before bed.
  Interventions: Drug: Bepotastine besilate
- ketotifen fumarate (Active Comparator): Two TAU-284 5mg placebo tablets and one ketotifen fumarate dry syrup 1g will be taken orally twice a day, once after breakfast and once before bed.
  Interventions: Drug: ketotifen fumarate

INTERVENTIONS:
Drug: Bepotastine besilate — Two TAU-284 5mg tablets and one ketotifen fumarate dry syrup 1g placebo will be taken orally twice a day
  Other Names: TALION 5mg tablets
  Arms: TAU-284
Drug: ketotifen fumarate — Two TAU-284 5 mg placebo tablets and one ketotifen fumarate dry syrup 1g will be taken orally twice a day
  Other Names: ketotifen fumarate dry syrup
  Arms: ketotifen fumarate

SUMMARY:
The objective of this study is to verify the non-inferiority of TAU-284 to ketotifen fumarate dry syrup in the change in the severity of pruritus after the treatment period.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-group comparative study to demonstrate the noninferiority of TAU-284 to ketotifen fumarate in pediatric patients with atopic dermatitis, as assessed by the primary endpoint of the change from baseline in pruritus score after 2-week treatment with TAU-284 (20 mg/day) or ketotifen fumarate dry syrup (2 g/day); and to investigate the safety, and plasma concentrations of TAU-284.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 7 and 15 years
* Patients giving assent and whose legal guardian giving informed consent
* Outpatients
* Patients diagnosed as atopic dermatitis
* Patients who require the treatment with topical corticosteroid on areas other than face, head and neck
* Patients whose diaries can be properly maintained
* Patients who have 2 grades or more pruritus score

Exclusion Criteria:

* Patients with bronchial asthma who require concomitant use of the corticosteroid
* Patients who have been undergoing specific desensitization therapy or nonspecific immunomodulation therapy or phototherapy
* Patients with current or previous history of drug hypersensitivity
* Patients who have been treated with Bepotastine besilate in the past
* Patients who have; a skin infection, or with zooparasite such as scabies and pediculosis; eczematous otitis externa with perforation in the eardrum; dermal ulcer, or profound heat burn or frostbite of the severity higher than the grade 2; on areas where topical corticosteroid is applied
* Patients who have spastic disease such as epilepsy
* Patients who concurrently have renal function abnormalities that may cause safety problems
* Patients who do not give consent to use birth control
* Pregnant patients, at risk of pregnancy or breastfeeding
* Patients who had participated in any clinical trial in the last 12 weeks

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MAKOTO KAWASHIMA, Study Director — Tokyo Women's Medical University
Locations (1):
- Medical Corporation Kojinkai Asanuma Dermatology Clinic, Hokkaido, Japan

REFERENCES:
- [Result] Kawashima M; Ichimura M; Yano K; Susuta Y; Izaki H. Phase III study of bepotastine besilate in children with atopic dermatitis -A randomized, double-blind, parallel-group, comparative study with ketotifen fumarate dry syrup- Rinsho iyaku 2015 Mar;31(3):235-251

RESULTS

PARTICIPANT FLOW:
Groups:
- TAU-284: TAU-284 10mg twice daily for 2 weeks
- Ketotifen Fumarate: Ketotifen fumarate dry syrup 1g twice daily for 2 weeks
Period: Overall Study
Arm/Group | TAU-284 | Ketotifen Fumarate
Started | 151 | 152
Completed | 149 | 150
Not Completed | 2 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAU-284 | Ketotifen Fumarate | Total
Number analyzed (Participants) | 151 | 152 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (2.3) | 10.4 (2.5) | 10.3 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 62 | 141
  Male | 72 | 90 | 162

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pruritus Score
Description: The pruritus symptoms score were rated on 5-point scale ranging from 0 (none) to 4 (severe).
Time Frame: Baseline and 2 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TAU-284 | Ketotifen Fumarate
Number analyzed (Participants) | 151 | 152
units on a scale | -0.669 (0.058) | -0.638 (0.058)

2. Secondary Outcome: Change From Baseline in Pruritus Score
Description: The pruritus symptoms score were rated on 5-point scale ranging from 0 (none) to 4 (severe).
Time Frame: Baseline and 1 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TAU-284 | Ketotifen Fumarate
Number analyzed (Participants) | 151 | 152
units on a scale | -0.425 (0.047) | -0.510 (0.047)

3. Secondary Outcome: Severity of Atopic Dermatitis at 2 Weeks (Change From Baseline)
Description: Severity score were rated on 5-point scale ranging from 0 (none) to 4 (severe).
Time Frame: Baseline and 2 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TAU-284 | Ketotifen Fumarate
Number analyzed (Participants) | 151 | 152
units on a scale | -0.8 (0.0) | -0.7 (0.0)

4. Secondary Outcome: Percentage of Participants With Patient Impression Score (Reporting Excellent or Very Well Improved in Pruritus)
Description: Patient impression score were rated on 5-point scale ranging from 0 to 4 (4 excellent, 3 very well, 2 well, 1fair, 0 poor).
Time Frame: Week 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAU-284 | Ketotifen Fumarate
Number analyzed (Participants) | 151 | 152
percentage of participants | 65.6 [57.4 to 73.1] | 65.1 [57.0 to 72.7]

ADVERSE EVENTS:
Arm/Group | TAU-284 | Ketotifen Fumarate
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/152
Other Adverse Events (participants affected / at risk) | 6/151 | 11/152
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAU-284 (N=151) | Ketotifen Fumarate (N=152)
Nasopharyngitis (Infections and infestations) | 3 | 6
Somnolence (Nervous system disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other